CLINICAL TRIAL: NCT05413551
Title: Point-of-care Pharmacogenomic Testing to Optimize Isoniazid Dosing for Tuberculosis Prevention
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Federal University of Mato Grosso (Other); Fiocruz Mato Grosso do Sul (Unknown)
Responsible Party: Principal Investigator, Jason Andrews, Associate Professor of Medicine, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 65808; 1R21AI172182-01 (NIH)
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-07

CONDITIONS: Tuberculosis Infection; Isoniazid Adverse Reaction
MeSH Terms: conditions — Latent Tuberculosis | interventions — Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Rapid acetylator (Experimental): Participants will receive 1 standard dose (Day 0), followed by 1 higher dose (Day 7), follow by 2 standard doses (Days 14 and 21).
  Interventions: Drug: Standard dose of isoniazid; Drug: High-dose isoniazid
- Intermediate acetylator (Active Comparator): Participants will receive 4 standard doses (Days 0, 7, 14 and 21).
  Interventions: Drug: Standard dose of isoniazid
- Slow acetylator (Experimental): Participants will receive 2 standard doses (Days 0 and 7), followed by 1 lower dose (Day 21), follow by 1 standard dose (Day 21).
  Interventions: Drug: Low-dose isoniazid; Drug: Standard dose of isoniazid

INTERVENTIONS:
Drug: Low-dose isoniazid — Pharmacogenomic-modified dose of isoniazid - 5 mg/kg oral tablet (maximum 300 mg)
  Arms: Slow acetylator
Drug: Standard dose of isoniazid — 15 mg/kg oral tablet (up to 900 mg)
Drug: High-dose isoniazid — Pharmacogenomic-modified dose of isoniazid - 25 mg/kg oral tablet (maximum 1500 mg)
  Arms: Rapid acetylator

SUMMARY:
This trial is designed to determine whether modifying the dose of isoniazid for individuals according to their n-acetyltransferase 2 (NAT2) genotype could increase the probability of achieving equivalence of area-under-the-curve.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for latent tuberculosis treatment by Brazil's national guidelines*
* provides written informed consent to participate in the study

Exclusion Criteria:

* Evidence of active tuberculosis or currently under evaluation for active tuberculosis
* Receiving drugs that interact with Rifapentine (e.g. methadone, warfarin)
* Known intolerance or hypersensitivity to isoniazid or rifapentine
* Prior treatment for active or latent tuberculosis > 14 days
* Close contact to isoniazid- or rifampicin-resistant tuberculosis (TB) case
* Neutropenia (absolute neutrophil count <1000 cells/mm3)
* Clinical diagnosis of active liver disease or alcohol dependence
* alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 times the upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Isoniazid plasma area-under-the-curve | 1, 2, 8, and 24 hours post-dose

SECONDARY OUTCOMES:
Maximum isoniazid concentration (Cmax) | 1, 2, 8, and 24 hours post-dose
Isoniazid concentration at 24 hours | 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Jason R Andrews, MD, Principal Investigator — Stanford University
Locations (1):
- Federal University of Mato Grosso do Sul, Campo Grande, Mato Grosso do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
We will make the study protocol, statistical analysis plan, informed consent form and report available. We will make a de-identified dataset available.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Verma R, Patil S, Zhang N, Moreira FMF, Vitorio MT, Santos ADS, Wallace E, Gnanashanmugam D, Persing DH, Savic RM, Croda J, Andrews JR. A Rapid Pharmacogenomic Assay to Detect NAT2 Polymorphisms and Guide Isoniazid Dosing for Tuberculosis Treatment. Am J Respir Crit Care Med. 2021 Dec 1;204(11):1317-1326. doi: 10.1164/rccm.202103-0564OC. PMID 34375564